CLINICAL TRIAL: NCT04635566
Title: Pharmacological Enhancement for Nocturnal Incontinence in Orthotopic Bladder Substitute. A Randomised Controlled Trial
Brief Title: Pharmacological Enhancement for Nocturnal Incontinence in Orthotopic Bladder Substitute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NE-OBS
Record Dates: First submitted 2020-11-14; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Incontinence; Urinary Incontinence; Urinary Bladder Cancer
Keywords: Incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder Neoplasms | interventions — mebeverine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mebeverine (Active Comparator): Mebeverine 200 mg sustained-release (Coloverine® SR, Chemipharm pharmaceutical, Egypt) one time/day at the evening.
  Interventions: Drug: mebeverine 200 mg sustained-release (Coloverine® SR, Chemipharm pharmaceutical, Egypt) one time/day at the evening.
- Placebo (Placebo Comparator): Placebo one time/day at the evening.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mebeverine 200 mg sustained-release (Coloverine® SR, Chemipharm pharmaceutical, Egypt) one time/day at the evening. — mebeverine 200 mg sustained-release (Coloverine® SR, Chemipharm pharmaceutical, Egypt) one time/day at the evening. 200 mg sustained-release (Coloverine® SR, Chemipharm pharmaceutical, Egypt) one time/day at the evening.
  Other Names: Coloverine® SR
  Arms: Mebeverine
Drug: Placebo — Placebo one time/day at the evening.
  Arms: Placebo

SUMMARY:
In this randomised trial, we hypothesised that mebeverine could enhance nocturnal continenece of Orthotopic Bladder Substitute (OBS) patients by decreasing the frequency and reduce maximum amplitude of uninhibited contractions of OBS ileum, and consequently it would increase the OBS capacity

ELIGIBILITY:
Inclusion Criteria:

* nocturnal enuresis

Exclusion Criteria:

* daytime incontinence
* Orthotopic Bladder Substitute (OBS) reconstruction surgery ≤2 years
* chronic kidney disease
* local tumor recurrence
* adjuvant chemotherapy and/or radiotherapy
* chronic retention requiring use of clean intermittent catheterization or indwelling urethral catheterization
* suspected or known narrow-angle glaucoma
* sensitivity to mebeverine.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients
Enrollment: 120 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
assess the 3-months nocturnal continence rate | 3 months
  comparing Urinary function domain from the bladder cancer index (BCI) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt